CLINICAL TRIAL: NCT03288155
Title: A Study to Determine Whether the Daily Consumption of Flavonoid-rich Pure Cocoa Can Reduce Fatigue in People With Parkinson's (PD)
Brief Title: Can a Flavonoid-rich Pure Cocoa Reduce Fatigue in People With Parkinson's (PD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Collaborators: European Parkinson Therapy Centre (Unknown)
Responsible Party: Principal Investigator, Shelly Coe, Principal investigator, Oxford Brookes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OxfordBU
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Parkinson Disease; Fatigue
Keywords: Parkinson's; Fatigue; Flavonoid; Cocoa
MeSH Terms: conditions — Parkinson Disease; Fatigue | interventions — Chocolate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind randomized controlled feasibility trial with assessors and participant blinded to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flavonoid rich cocoa (Experimental): Dark cocoa beverage rich in flavonoids
  Interventions: Dietary Supplement: Cocoa
- Low flavonoid cocoa (Placebo Comparator): A control cocoa beverage low inn flavonoids
  Interventions: Dietary Supplement: Cocoa

INTERVENTIONS:
Dietary Supplement: Cocoa — Participants will receive either a high flavonoid cocoa or a low flavonoid placebo cocoa.

SUMMARY:
This study determines to evaluate the effectiveness of the daily consumption of flavonoid-rich cocoa in the treatment of fatigue in Parkinson's patients. The participants were divided equally between the flavonoid-rich cocoa (device) and control cocoa groups. The participant will engage in a six day trial, with measures taken at Day 1 and Day 6.

DETAILED DESCRIPTION:
Many pwPD have expressed their interest in dietary therapies to manage their symptoms; however scientific evidence for these therapies is lacking. Flavonoids, plant compounds found in certain foods, may have the ability to improve fatigue. However, to date, no well-designed intervention studies assessing the role of flavonoid consumption for fatigue management in pwPD have been performed.

The aim of this project is to undertake a feasibility preliminary study to determine whether flavonoid-rich cocoa has the potential to improve fatigue in pwPD in order to inform a follow on trial. Participants will be recruited from the European Parkinson Therapy Centre (EPTC) and will be those about to enrol onto the 6 day program. They will be required to consume a cocoa drink each morning for 6 days. They will have measures taken including fatigue measures using visual rating scales, walking tests and several questionnaires will be administered during this time.

Aims:

The hypothesis is that the consumption of a flavonoid-rich pure cocoa beverage will reduce fatigue in pwPD. The aim of this study is to determine the feasibility of a trial to evaluate this proposal.

Design:

This is a randomised double-blind placebo controlled feasibility study in which 20 (+ potentially 20 more if adherence is acceptable and recruitment is progressing as expected) pwPD will be recruited from the European Parkinson Therapy Centre (EPTC), Italy.

Intervention:

A 6 day nutrition intervention period, with a total of 2 assessments (baseline and day 6) where outcome measures will be assessed.

Population:

20 men and women with a diagnosis of PD and who are over 18 years of age. There will be 10 participants in each trial arm.

Outcome Measures:

In order to assess benefits, a range of outcomes will be obtained. Outcome measures include:

Levels of physical activity: wearable activity monitors (worn like a watch)

Dietary patterns: 2-24 hour dietary record

Fatigue levels: Fatigue Severity Scale (FSS) and during the intervention the numerical rating scale (NRS) 3 times daily

Fatigability: performance on 6 minute walk test (physical) and AMIPB cognitive test

Health descriptives: basic health questionnaire, Euroqol (EQ5DVAS), SF36 Health survey, Unified Parkinson's Disease Rating Scale non motor symptoms (UPDRSNMS), routinely administered to the centre by Trescore Hospital.

Duration and follow-up:

Participants will be consented by a trained researcher at the Centre and, if successfully pass the eligibility check will be enrolled into the study. Staff at the Centre will be trained on taking consent by researchers at OBU. Once a participant is enrolled, a baseline assessment (Assessment 1) will be conducted at day 1. Immediately following completion of Assessment 1, participants will be randomly allocated to either the high flavonoid intervention group or the control group, and intervention delivery will begin immediately after allocation. They will be reassessed at day 6. Those in the control group will follow the same procedure, the only difference being that they receive the low flavonoid drink. Alex Reed and the EPTC will inform participant GPs about their involvement in the study.

ELIGIBILITY:
Inclusion Criteria

* 18 years + with a clinical diagnosis of Parkinson's disease
* Sufficient mental capacity to consent
* Score of 1-2 on Hoehn and Yahr scale

Exclusion Criteria

* Change in medication before the previous week of the trial and/ or an expected change during
* Known psychiatric disorder (clinically diagnosed)
* Contraindications tolerating the cocoa drink
* Other conditions that may be associated with fatigue, e.g. Anaemia
* Condition affecting the central nervous system other than Parkinson's disease (however migraine is allowed)
* Pregnant or lactating
* Objection to contacting their GP and neurologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Fatigue Numerical Scale (FNS) | Change from Baseline to Day 6
  The FFS measures the fatigue of an individual at set times throughout the day

SECONDARY OUTCOMES:
Adult Memory and Information Processing Battery (AMIPB) | Measurements taken at baseline and Day 6
  The AIMPB test is taken after a fasted night, provided unseen to the participant. The participant must circle the second highest number out of five. There are ten lines of numbers. The test is timed.
6-Minute Walking Test | Measurements taken at baseline and Day 6
  The 6-minute walking test measures the participants' physical competency. It is taken after the AIMPB (on a fasted stomach). The participant must walk around a set course, of 13 metres, which is timed.
Dietary Recall | Measurements taken at baseline and Day 6
  The dietary recall is taken to ensure any extraneous factors, potentially affecting the severity of Parkinson's symptoms or fatigue. The dietary recall is taken on the first (Day 1) and last day (Day 6) of the trial. The participants are not notified of the dietary recall commencement dates, to ensure they do not change their natural eating habits.
Accelerometer | Measurements continuously taken from baseline to Day 6
  The accelerometer measures the amount of activity expended by the participant during the duration of the trial (Day 1 to day 6). This is used to help distinguish variations between the FNS results, as well as fatigue related to physical exertion.
Final Evaluation Interview | Taken at day 6
  This questionnaire is to discover views from the participant upon the cessation of the trial. Including whether the participant will continue to drink the cocoa.

CONTACTS AND LOCATIONS:
Overall Officials: Shelly A Coe, PhD, Principal Investigator — Oxford Brookes Univeristy; Alex Reed, Study Director — European Parkinson Therapy Centre
Locations (1):
- European Parkinson Therapy Centre, Boario, Terme, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data would be anonymised and potentially available for public use

REFERENCES:
- [Derived] Coe S, Andreoli D, George M, Collett J, Reed A, Cossington J, Izadi H, Dixon A, Mansoubi M, Dawes H. A feasibility study to determine whether the daily consumption of flavonoid-rich pure cocoa has the potential to reduce fatigue and fatigability in people with Parkinson's (pwP). Clin Nutr ESPEN. 2022 Apr;48:68-73. doi: 10.1016/j.clnesp.2022.01.023. Epub 2022 Jan 31. PMID 35331536